CLINICAL TRIAL: NCT00202566
Title: Evaluation of the Anti-anginal Efficacy and Safety of Oral Administration of Ivabradine Compared to Placebo on Top of Background Therapy With Atenolol in Patients With Stable Angina Pectoris. A Four-month Randomised Double-blind, Parallel Group International Multicentre Study.
Brief Title: Efficacy and Safety of Ivabradine on Top of Atenolol in Stable Angina Pectoris
Acronym: ASSOCIATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CL3-16257-057
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Ivabradine

INTERVENTIONS:
Drug: Ivabradine

SUMMARY:
To test whether ivabradine when given in combination with atenolol is able to improve the exercise tolerance of patients with stable angina pectoris

ELIGIBILITY:
Inclusion Criteria:

* Chronic stable angina pectoris
* Documented coronary artery disease
* Previous treatment with atenolol or other beta-blocker agent
* Exercise tolerance test positivity and stability

Exclusion Criteria:

* Heart rate < 60 bpm
* Congestive heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2005-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Improvement between baseline and end of treatment of the treadmill exercise tolerance test

SECONDARY OUTCOMES:
Rate pressure product
Clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Tardif, Pr, Study Chair — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Result] Tardif JC, Ponikowski P, Kahan T; ASSOCIATE Study Investigators. Efficacy of the I(f) current inhibitor ivabradine in patients with chronic stable angina receiving beta-blocker therapy: a 4-month, randomized, placebo-controlled trial. Eur Heart J. 2009 Mar;30(5):540-8. doi: 10.1093/eurheartj/ehn571. Epub 2009 Jan 9. PMID 19136486